CLINICAL TRIAL: NCT06222411
Title: Does Leadership Training Affect Physician Career Satisfaction?
Brief Title: Leadership Training Affect Physician Career Satisfaction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 042.MBSI.2023.D
Record Dates: First submitted 2024-01-16; First posted 2024-01-24 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Leadership; Personality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physicians in Methodist Health System (MHS) (Other): All Current physicians who are older than 18 years of age who are literate in English
  Interventions: Other: evaluate the impact of organizational interventions for physician development on wellbeing

INTERVENTIONS:
Other: evaluate the impact of organizational interventions for physician development on wellbeing — There is an increasing demand for healthcare organizations and hospitals to address factors contributing to stress and burnout as well as provide effective solutions at an organizational level

SUMMARY:
The aim of the study is to evaluate the impact of organizational interventions for physician development on wellbeing, and investigate wellbeing and other characteristics of physicians with and without formal leadership roles.

DETAILED DESCRIPTION:
1. Compare the incidence of job satisfaction, stress, and burnout overall between physicians who have undergone some sort of leadership training and those who have not.
2. Compare the incidence of job satisfaction, stress, and burnout overall between physicians with and without formal leadership roles.
3. Determine additional factors associated with job satisfaction, stress, and burnout levels.
4. Evaluate intrinsic and extrinsic motivating factors associated with physicians currently in formal leadership roles and those interested in pursuing formal leadership roles in the future.
5. Determine whether more satisfied physicians seek leadership roles or whether seeking leadership roles leads to greater satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years
* Be a current licensed physician practicing at Methodist Health System( MHS )
* Literate in English
* Able and willing to provide consent

Exclusion Criteria:

* <18 years of age
* Not a current licensed physician at MHS
* Illiterate in English
* Unable or unwilling to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of incidence | 3 weeks
  Compare the incidence of job satisfaction, stress, and burnout overall between physicians who have undergone some sort of leadership training and those who have not.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Institute at Methodist Health System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No